CLINICAL TRIAL: NCT06300710
Title: Outcome of Cardiopulmonary Resuscitation in Tertiary Level PICU and Associated Risk Factors
Brief Title: Outcomes and Risk Factors of CPR in PICU
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Hamed Khalaf Ahmed, Principal investigator, Assiut University
Other Study IDs: CPR in PICU
Record Dates: First submitted 2024-02-21; First posted 2024-03-08 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-03

CONDITIONS: Cardio Respiratory Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To detect the frequency and the underlying causes of cardiopulmonary arrest .
2. To detect outcome of CPR
3. To identify the associated risk factors for the different outcomes after CPR among those patients

DETAILED DESCRIPTION:
Cardiac arrest (CA) is uncommon in children, and the epidemiology of pediatric CA is different from adults. CA Is a critical cause of death in children in the hospital especially in the pediatric Intensive care unit (PICU). CA Is reported in 2-6% of children in the PICU, which is much higher than out-of-hospital arrest (about 8 to 20 annual cases per 100,000 pediatric population .

Previous studies reported that return of spontaneous circulation (ROSC) after cardiopulmonary Resuscitation (CPR) for in-hospital CA (IHCA) is about half of these patients, and ∼30% survived to hospital discharge Previous studies had analyzed the cause and prognostic factors associated with outcomes after IHCA, which included the Initial rhythm, duration of CA and CPR, the underlying disease, and where the event attacked .

Patients in PICU are more likely to develop CA because they are more critically ill. Information on factors associated with prognosis of in-PICU CA can promote Improvement in PICU care, which means improving survival with good neurologic outcomes .

Analyzing the epidemiological variables and risk/prognostic factors of in-PICU CA is of great Importance in developing the better therapeutic strategy and deciding appropriate preventive Measure .

Probability of death on admission and a longer length Of stay in the PICU were associated with increased odds of receiving CPR. Children admitted with cardiac conditions were at significantly higher risk of receiving CPR in the PICU Compared with those Admitted with noncardiac primary diagnosis. The risk Of receiving CPR was significantly associated with age, History of preadmission CPR, also, Electrolyte Imbalances and Multi-organ Dysfunction increase risk of receiving CPR in PICU .

ELIGIBILITY:
Inclusion Criteria:

* Including Children aged 1 month to 18 years who received at least 1 minute of CPR

Exclusion Criteria:

* Exclusion of 1-Children aged below1 month and older than 18 years .
* terminal disease patients, such as malignancy

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children aged from 1 month to 18 years who suffered in-PICU CA between March 2024 to February 2025 will be included. Cardiopulmonary arrest was defined as the presence of unresponsiveness, apnea, absence of signs of life, and absence of a palpable central pulse or bradycardia of <60 bpm with poor perfusion in infants, requiring external cardiac compressions and assisted ventilation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
incidence of cardiac arrest and survival to discharge from the PICU (dead versus alive) | 1 year
  (dead versus alive)

SECONDARY OUTCOMES:
Rate of risk factors associated with outcome of CPR | 1 year
  Rate of the risk factors associated with the outcome of CPR.

REFERENCES:
- [Background] Lee EP, Chan OW, Lin JJ, Hsia SH, Wu HP. Risk Factors and Neurologic Outcomes Associated With Resuscitation in the Pediatric Intensive Care Unit. Front Pediatr. 2022 Apr 4;10:834746. doi: 10.3389/fped.2022.834746. eCollection 2022. PMID 35444968
- [Background] Choi J, Choi AY, Park E, Moon S, Son MH, Cho J. Trends in Incidences and Survival Rates in Pediatric In-Hospital Cardiopulmonary Resuscitation: A Korean Population-Based Study. J Am Heart Assoc. 2023 Feb 7;12(3):e028171. doi: 10.1161/JAHA.122.028171. Epub 2023 Jan 25. PMID 36695322
- [Background] Perkins GD, Jacobs IG, Nadkarni VM, Berg RA, Bhanji F, Biarent D, Bossaert LL, Brett SJ, Chamberlain D, de Caen AR, Deakin CD, Finn JC, Grasner JT, Hazinski MF, Iwami T, Koster RW, Lim SH, Huei-Ming Ma M, McNally BF, Morley PT, Morrison LJ, Monsieurs KG, Montgomery W, Nichol G, Okada K, Eng Hock Ong M, Travers AH, Nolan JP; Utstein Collaborators. Cardiac arrest and cardiopulmonary resuscitation outcome reports: update of the Utstein Resuscitation Registry Templates for Out-of-Hospital Cardiac Arrest: a statement for healthcare professionals from a task force of the International Liaison Committee on Resuscitation (American Heart Association, European Resuscitation Council, Australian and New Zealand Council on Resuscitation, Heart and Stroke Foundation of Canada, InterAmerican Heart Foundation, Resuscitation Council of Southern Africa, Resuscitation Council of Asia); and the American Heart Association Emergency Cardiovascular Care Committee and the Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation. Circulation. 2015 Sep 29;132(13):1286-300. doi: 10.1161/CIR.0000000000000144. Epub 2014 Nov 11. PMID 25391522
- [Background] Kuisma M, Suominen P, Korpela R. Paediatric out-of-hospital cardiac arrests--epidemiology and outcome. Resuscitation. 1995 Oct;30(2):141-50. doi: 10.1016/0300-9572(95)00888-z. PMID 8560103
- [Background] Reis AG, Nadkarni V, Perondi MB, Grisi S, Berg RA. A prospective investigation into the epidemiology of in-hospital pediatric cardiopulmonary resuscitation using the international Utstein reporting style. Pediatrics. 2002 Feb;109(2):200-9. doi: 10.1542/peds.109.2.200. PMID 11826196